CLINICAL TRIAL: NCT07311148
Title: A Phase Ⅱ, Randomized, Observer-blinded, Parallel-Controlled Clinical Trial to Assess the Immunogenicity and Safety of the Recombinant Zoster Vaccine, LYB004 in Adults Aged 40 Years and Older
Brief Title: A Immunogenicity and Safety Trial of the Recombinant Zoster Vaccine （CHO Cell）, LYB004 in Adults Aged 40 Years and Older
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LYB004/CT-CHN-201
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Herpes Zoster (HZ); Shingles; VZV; Recombinant Zoster Vaccine
Keywords: herpes zoster; varicella-zoster virus; Virus-like particles; Recombinant protein vaccine; Glycoprotein E
MeSH Terms: conditions — Herpes Zoster; Chickenpox | interventions — Antigens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low dose antigen and low dose adjuvant of LYB004 (Experimental): Participants aged 40 years and older will be vaccinated with 2 doses of LYB004 (low dose antigen and low dose adjuvant) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Low dose antigen and low dose adjuvant of LYB004
- Low dose antigen and high dose adjuvant of LYB004 (Experimental): Participants aged 40 years and older will be vaccinated with 2 doses of LYB004 (low dose antigen and high dose adjuvant ) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Low dose antigen and high dose adjuvant of LYB004
- High dose antigen and low dose adjuvant of LYB004 (Experimental): Participants aged 40 years and older will be vaccinated with 2 doses of LYB004 (high dose antigen and low dose adjuvant) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: High dose antigen and low dose adjuvant of LYB004
- High dose antigen and high dose adjuvant of LYB004 (Experimental): Participants aged 40 years and older will be vaccinated with 2 doses of LYB004 (high dose antigen and high dose adjuvant) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: High dose antigen and high dose adjuvant of LYB004
- Placebo (Placebo Comparator): Participants aged 40 years and older will be vaccinated with 2 doses of placebo on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Placebo
- Positive control (Active Comparator): Participants aged 50 years and older will be vaccinated with 2 doses of Shingrix® on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Positive control

INTERVENTIONS:
Biological: Low dose antigen and low dose adjuvant of LYB004 — 0.5 mL per dose, containing 25 μg VZV-gEM adjuvanted with A01C.
  Arms: Low dose antigen and low dose adjuvant of LYB004
Biological: Low dose antigen and high dose adjuvant of LYB004 — 0.5 mL per dose, containing 25 μg VZV-gEM adjuvanted with A01B.
  Arms: Low dose antigen and high dose adjuvant of LYB004
Biological: High dose antigen and low dose adjuvant of LYB004 — 0.5 mL per dose, containing 50 μg VZV-gEM adjuvanted with A01C.
  Arms: High dose antigen and low dose adjuvant of LYB004
Biological: High dose antigen and high dose adjuvant of LYB004 — 0.5 mL per dose, containing 50 μg VZV-gEM adjuvanted with A01B.
  Arms: High dose antigen and high dose adjuvant of LYB004
Biological: Placebo — 0.5 mL per dose, without antigen and adjuvant.
  Arms: Placebo
Biological: Positive control — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with AS01B.
  Arms: Positive control

SUMMARY:
This phase 2 study in China will evaluate the immunogenicity and safety of the Recombinant Zoster Vaccine, LYB004 in adults aged 40 years and older.

DETAILED DESCRIPTION:
A randomized, observer-blinded, parallel-controlled trial will be conducted to observe the immunogenicity and safety of LYB004 in adults aged 40 years and older. A total of 840 participants aged 40 years and older will be enrolled. Four formulations of LYB004 will be provided: two dose levels of antigen and two dose levels of adjuvant. Participants aged 40-49 years old will randomly receive four investigational vaccines and the placebo in a 2:2:2:2:1 ratio. Participants aged 50 years and older will randomly receive four investigational vaccines, positive control and the placebo in a 2:2:2:2:2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Residents aged 40 years and older (at the time of screening), regardless of gender;
2. Participants can provide valid identification, voluntarily agree to participate in the study, and sign the Informed Consent Form;
3. Participants are able to attend all planned follow-up visits and comply with the protocol requirements;
4. Females of childbearing potential should use effective contraceptive measures one month before enrollment; females of childbearing potential (excluding those who have undergone tubal ligation, bilateral oophorectomy, or hysterectomy) and male participants should practice effective contraception and avoid pregnancy plans, as well as sperm or egg donation plans from the time of enrollment until 6 months after the full course of vaccination. Effective contraceptive methods include oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release local contraceptives, contraceptive patches, intrauterine devices, sterilization, abstinence, condoms, diaphragms, cervical caps, etc.

Exclusion Criteria:

1. Axillary temperature ≥ 37.0°C;
2. History of herpes zoster before vaccination with the investigational vaccine;
3. Previous vaccination against HZ or varicella;
4. Has had close contact with patients with varicella/herpes zoster within 6 months before vaccination with the investigational vaccine;
5. Has received any vaccine within 14 days before vaccination, or have received a live vaccine within 28 days;
6. Those who have received blood or blood-related products, including immunoglobulins, within 3 months before the first dose of vaccination, or have planned to use them during the study period;
7. Individual with the following diseases: ① Have acute diseases or are in the acute exacerbation period of chronic diseases, or take antipyretic, analgesic, and anti-allergic drugs within 3 days before vaccination; ② Allergies to any component of the study vaccine, or have a history of severe allergic reactions to any vaccination; ③ History of convulsions, epilepsy, encephalopathy (such as congenital brain dysplasia, brain trauma, brain tumors, cerebral hemorrhage, cerebral infarction, brain infection, chemical poisoning, etc. causing brain nerve tissue damage, etc.) and mental illness, or a family history of mental illness; ④ Asplenia, or functional asplenia; ⑤Primary or secondary immunodeficiency, or diagnosed with congenital or acquired immunodeficiency, human immunodeficiency virus infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune diseases; ⑥ Chronic administration (≥14 consecutive days) of glucocorticoid (reference value for dose: ≥ 2mg/kg/day or ≥ 20mg/day prednisone or equivalent) or other immunosuppressive agents within the past 3 months, with the exception of inhaled or topical steroids, or short-term use (<14 consecutive days) of oral corticosteroids; ⑦ Severe cardiovascular diseases (pulmonary heart disease, pulmonary edema, etc.), severe liver and kidney diseases, complicated diabetes; ⑧ History of thrombocytopenia or other coagulation disorders that may contraindicate intramuscular injection;⑨Severe hypertension that cannot be controlled by medication (on-site measurement: systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg);
8. Those tested positive for antibodies to the Human Immunodeficiency Virus (HIV) at screening.;
9. History of long-term alcohol abuse and/or drug abuse;
10. Individual who is currently participating in other research or unregistered product (drugs, vaccines, or devices, etc.) clinical studies, or plan to participate in other clinical studies before the end of this clinical study;
11. Exclusion criteria for specific populations: lactating or pregnant women during the clinical research period, or women of childbearing age with a positive pregnancy test before vaccination;
12. Other conditions that may impact the subject's safety or influence the assessment of vaccine response, as determined by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The geometric mean concentration (GMC) of anti-glycoprotein E (gE) antibody | 30 days after second vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA).
The geometric mean titer (GMT) of anti-VZV antibody | 30 days after second vaccination
  Measured by fluorescent antibody to the membrane antigen (FAMA).

SECONDARY OUTCOMES:
Occurrence of immediate adverse events | Within 30 minutes after each vaccination
  The incidence and severity of any adverse events (AEs) within 30 minutes after each vaccination
Incidence of solicited AE | Within 0-7 days after each vaccination
  Occurrence and severity of solicited local injection site reactions for 7 days (Day 0-Day 7) following each vaccination. (i.e., pain, redness, swelling).
  Occurrence and severity of solicited systemic reactions for 7 days (Day 0-Day 7) following each vaccination. (i.e., myalgia, fatigue, headache, chills, fever).
Incidence of unsolicited AEs | Within 30 days after each vaccination
  The incidence and severity of any unsolicited AEs, including all AEs, except solicited AEs reported Days 0~30 after the study intervention. vaccination
Occurrence of serious adverse events (SAEs) and adverse events of special interests (AESIs) | From the first vaccination up to 12 months after the second vaccination
  The incidence of any serious adverse events (SAEs) and adverse events of special interest (AESIs) from the first vaccination up to 12 months after the second vaccination
The geometric mean titer (GMT) of anti-VZV antibody | 60 days after first vaccination, 6 months and 12 months after second vaccination
  Measured by fluorescent antibody to the membrane antigen (FAMA).
The geometric mean concentration (GMC) of anti-glycoprotein E (gE) antibody | 60 days after first vaccination, 6 months and 12 months after second vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA).
The seroconversion rate of anti-Varicella Zoster Virus (VZV) antibody | 60 days after first vaccination, 30 days, 6 months and 12 months after second vaccination
  Seroconversion refers to at least a 4-fold increase in the anti-Varicella Zoster Virus (VZV) antibody titer at the endpoint as compared to the prevaccination titer if prevaccination titer is above the lower limit of quantification (LLOQ) or a 4-fold increase at the endpoint as compared to LLOQ value if prevaccination concentration is lower than LLOQ.
The seroconversion rate of anti-glycoprotein E (gE) antibody | 60 days after first vaccination, 30 days, 6 months and 12 months after second vaccination
  Seroconversion refers to at least a 4-fold increase in the anti-glycoprotein E (gE) antibody concentration at the endpoint as compared to the prevaccination concentration if prevaccination concentration is above the lower limit of quantification (LLOQ) or a 4-fold increase at the endpoint as compared to LLOQ value if prevaccination concentration is lower than LLOQ.
The geometric mean fold rise (GMFR) of anti-VZV antibody | 60 days after first vaccination, 30 days, 6 months and 12 months after second vaccination
  Change from prevaccination in geometric mean fold rise of anti-VZV antibody titer.
The GMFR of anti-gE antibody | 60 days after first vaccination, 30 days, 6 months and 12 months after second vaccination
  Change from prevaccination in geometric mean fold rise of anti-gE antibody concentration.
Frequencies of CD4+ T cells secreting at least two of gE specific activation markers (IFN-γ, IL-2, TNF-α, CD40L) per 10^6 CD4+ T cells, and the cell mediated immunity (CMI) response rates at timepoints during the study | 30 days, 6 months and 12 months after second vaccination
  The frequencies of CD4+ T cells secreting at least two of gE specific activation markers (IFN-γ, IL-2, TNF-α, CD40L) per 10^6 CD4+ T cells, and the cell mediated immunity (CMI) response rates at 30 days and 6 months after second vaccination.
Frequencies of CD8+ T cells secreting at least two of gE specific activation markers (IFN-γ, IL-2, TNF-α, CD40L) per 10^6 CD8+ T cells, and the cell mediated immunity (CMI) response rates at timepoints during the study | 30 days, 6 months and 12 months after second vaccination
  The frequencies of CD8+ T cells secreting at least two of gE specific activation markers (IFN-γ, IL-2, TNF-α, CD40L) per 10^6 CD8+ T cells, and the cell mediated immunity (CMI) response rates at 30 days after first vaccination, 30 days and 6 months after second vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hengnan County Center for Disease Control and Prevention, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided